CLINICAL TRIAL: NCT01380964
Title: Research of Biomarkers for Disease Diagnosis, Disease Monitoring and Therapeutic Treatment Response in Duchenne Muscular Dystrophy Patients
Brief Title: Research of Biomarkers in Duchenne Muscular Dystrophy Patients
Acronym: IBISD
Status: Completed | Type: Observational
Sponsor: Genethon (Other)
Collaborators: Institute of Myology (Other)
Responsible Party: Sponsor
Other Study IDs: GEE006.10
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
Keywords: Duchenne Muscular Dystrophy; biomarkers; transcriptomics; mironics; proteomics
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, serum, t lymphocytes, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- DMD patients: DMD Patients
- Control patients: Control patients

SUMMARY:
The purpose of this study is to identify potential biomarkers for the diagnosis, disease progression assessment and response to treatment in patients with Duchenne Muscular Dystrophy.

ELIGIBILITY:
Inclusion Criteria:

* FOR PATIENTS:
* Diagnosis of DMD confirmed by genetic testing
* Age over 3 years
* Weight over 15 kg
* Informed consent signed
* FOR CONTROLS:
* Age over 3 years
* Male gender
* Weight over 15 kg
* Subjects with national health insurance coverage
* Informed consent signed
* Nonacute or chronic muscular, allergic, infectious, endocrine or inflammatory disorder in the 3 weeks preceding inclusion

Exclusion Criteria:

* FOR PATIENTS:
* Concomitant chronic or acute muscular, endocrine, infectious, allergic or inflammatory disorder in the three weeks preceding the blood test
* Intake of medicines other than angiotensin-converting enzyme inhibitors, beta blockers, dietary supplements, vitamins, alendronate and methylphenidate. Steroids (and medicines prescribed with them such as calcium supplements and proton pump inhibitors) will be discussed
* Mental retardation or autism
* Vaccination or treatment with immunoglobulins within the three months preceding inclusion
* FOR CONTROLS:
* Concomitant chronic or acute muscular, neurological (including mental retardation and autism), infectious or inflammatory disorder in the three weeks preceding the blood test
* Vaccination or treatment with immunoglobulins within the three months preceding inclusion

Ages: 3 Years to 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: patients with Duchenne Muscular Dystrophy controls (healthy or patients with a non-related disease)
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2011-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
IBiSD aims to identify and validate new and disease-specific biomarkers. | End of study
  This study will establish the relevance of urinary and blood biomarkers for the diagnosis, follow-up and assessment of treatment response in patients with DMD (IBiSD1, 2 and 4). IBiSD will also attempt to establish the seroprevalence to the different strains of AAV in patients with DMD (IBiSD3).

CONTACTS AND LOCATIONS:
Overall Officials: Laurent SERVAIS, MD, Principal Investigator — Myology Institute
Locations (1):
- Institute of Myology, Paris, France